CLINICAL TRIAL: NCT05003661
Title: The Effects of the Parents' Voice to Reduce the Heel Puncture Pain in High-Risk Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: YM109151F
Record Dates: First submitted 2021-07-18; First posted 2021-08-12 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Pain
Keywords: Parents voice; Heel Puncture; Neonatal pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mother's voice (Experimental): Neonates receive the intervention that recording of mother's voice of reading children's book. And the pain of high-risk newborns was measured with the Heartbeat, Respiration, SPO2 and Neonatal Infant Pain Scale (NIPS) in three minutes before the heel puncture, during the puncture, and the first, fifth and tenth minutes after the puncture.
  Interventions: Behavioral: Parents' Voice
- Father's voice (Experimental): Neonates receive the intervention that recording of father's voice of reading children's book. And the pain of high-risk newborns was measured with the Heartbeat, Respiration, SPO2 and Neonatal Infant Pain Scale (NIPS) in three minutes before the heel puncture, during the puncture, and the first, fifth and tenth minutes after the puncture.
  Interventions: Behavioral: Parents' Voice
- control group (No Intervention): When the infants undergoing heel puncture procedure, the control group were under routine care. And the pain of high-risk newborns was measured with the Heartbeat, Respiration, SPO2 and Neonatal Infant Pain Scale (NIPS) in three minutes before the heel puncture, during the puncture, and the first, fifth and tenth minutes after the puncture.

INTERVENTIONS:
Behavioral: Parents' Voice — the intervention is recording of parents voice of reading children's book.
  Arms: Father's voice; Mother's voice

SUMMARY:
High-risk neonates are forced to be separated from their parents due to hospitalization, and clinical medical treatment often causes pain and physical stress in high-risk newborns. Many literatures have confirmed that the mother's voice is positively helpful to the physiology of high-risk newborns, but few studies have been conducted on the father's voice. However, the parenting process is not only a link between the mother-child relationship, but also the impact of parental voice on high-risk newborns infants. Parent roles are expecting. The purpose of this study is to explore the effectiveness of parental voice intervention in high-risk newborns' heel puncture in reducing pain, and to further compare the mother and father's voice characteristics to the analysis of the pain degree of high-risk newborns.

DETAILED DESCRIPTION:
This study is a kind of experimental research design. The subjects are 105 infants with gestational weeks of more than 32 weeks. Randomly allocated are divided into one group of 35 in control group and 35 in each experimental group. On the third day after the birth of the high-risk newborns infant, the heel puncture times is lasted three minutes before the heel puncture to ten minutes after the puncture. The control groups only received general routine care, while the two parental experimental groups received the intervention that recording of parents voice of reading children's book. In the three groups, the pain of high-risk newborns was measured with the Heartbeat, Respiration and Neonatal Infant Pain Scale (NIPS) in three minutes before the heel puncture, during the puncture, and the first, fifth and tenth minutes after the puncture. It is hoped that the results of this study can help high-risk newborns to reduce pain with non-drug measures, and understand the influence of different voice characteristics on the development of infants, so as to provide future care personnel assisting parental role expectation and reference of clinical care.

ELIGIBILITY:
Inclusion Criteria:

* High-risk newborns over 32 weeks of age.
* Those who want to receive blood film collection for newborn screening on the third day of birth.
* The incubator is used for care during the hospitalization.
* The mother or father of the research subject can participate in the test all the way.
* After explaining and reading the consent form, the parents of the research subjects agree to participate in the research and obtain written consent.

Exclusion Criteria:

* Apgar Score is still below 7 in the fifth minute.
* Being treated with a high-frequency positive pressure respirator.
* Suffering from congenital diseases including: ear canal malformation, cerebral palsy, Down's syndrome, congenital cyanotic heart disease.
* After the doctor's assessment, the patient should continue fasting due to the condition or restrict breastfeeding on demand.
* Instability of blood glucose after birth requires close monitoring of blood glucose, and has received more than three (including) heel puncture experiences.
* Birth injuries of the body due to the birth process, such as broken fetal head and broken collarbone.
* Are receiving medical treatment with sedatives.

Min Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-09-26 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Change in heart rate from 3rd minute before the heel puncture to 10th minute after the heel puncture | Measure the heart rate at 3rd minute before the heel puncture
  Measure the heart rate at 3rd minute before the heel puncture, during, and at 1st, 5th and 10th minutes after the heel puncture
Change in heart rate from 3rd minute before the heel puncture to 10th minute after the heel puncture | Measure the heart rate during the heel puncture
  Measure the heart rate at 3rd minute before the heel puncture, during, and at 1st, 5th and 10th minutes after the heel puncture.
Change in heart rate from 3rd minute before the heel puncture to 10th minute after the heel puncture | Measure the heart rate at 1st minute after the heel puncture
  Measure the heart rate at 3rd minute before the heel puncture, during, and at 1st, 5th and 10th minutes after the heel puncture
Change in heart rate from 3rd minute before the heel puncture to 10th minute after the heel puncture | Measure the heart rate at 5th minute after the heel puncture
  Measure the heart rate at 3rd minute before the heel puncture, during, and at 1st, 5th and 10th minutes after the heel puncture
Change in heart rate from 3rd minute before the heel puncture to 10th minute after the heel puncture | Measure the heart rate at 10th minute after the heel puncture
  Measure the heart rate at 3rd minute before the heel puncture, during, and at 1st, 5th and 10th minutes after the heel puncture
Change in respiratory rate from 3rd minute before the heel puncture to 10th minute after the heel puncture | Measure the respiratory rate at 3rd minute before the heel puncture
  Measure the respiratory rate at 3rd minute before the heel puncture, during, and at 1st, 5th and 10th minutes after the heel puncture
Change in respiratory rate from 3rd minute before the heel puncture to 10th minute after the heel puncture | Measure the respiratory rate during the heel puncture
  Measure the respiratory rate at 3rd minute before the heel puncture, during, and at 1st, 5th and 10th minutes after the heel puncture
Change in respiratory rate from 3rd minute before the heel puncture to 10th minute after the heel puncture | Measure the respiratory rate at 1st minute after the heel puncture
  Measure the respiratory rate at 3rd minute before the heel puncture, during, and at 1st, 5th and 10th minutes after the heel puncture
Change in respiratory rate from 3rd minute before the heel puncture to 10th minute after the heel puncture | Measure the respiratory rate at 5th minute after the heel puncture
  Measure the respiratory rate at 3rd minute before the heel puncture, during, and at 1st, 5th and 10th minutes after the heel puncture
Change in respiratory rate from 3rd minute before the heel puncture to 10th minute after the heel puncture | Measure the respiratory rate at 10th minute after the heel puncture
  Measure the respiratory rate at 3rd minute before the heel puncture, during, and at 1st, 5th and 10th minutes after the heel puncture
Change in oxygen saturation from 3rd minute before the heel puncture to 10th minute after the heel puncture | Measure the oxygen saturation at 3rd minute before the heel puncture
  Measure the oxygen saturation at 3rd minute before the heel puncture, during, and at 1st, 5th and 10th minutes after the heel puncture
Change in oxygen saturation from 3rd minute before the heel puncture to 10th minute after the heel puncture | Measure the oxygen saturation during the heel puncture
  Measure the oxygen saturation at 3rd minute before the heel puncture, during, and at 1st, 5th and 10th minutes after the heel puncture
Change in oxygen saturation from 3rd minute before the heel puncture to 10th minute after the heel puncture | Measure the oxygen saturation at 1st minute after the heel puncture
  Measure the oxygen saturation at 3rd minute before the heel puncture, during, and at 1st, 5th and 10th minutes after the heel puncture
Change in oxygen saturation from 3rd minute before the heel puncture to 10th minute after the heel puncture | Measure the oxygen saturation at 5th minute after the heel puncture
  Measure the oxygen saturation at 3rd minute before the heel puncture, during, and at 1st, 5th and 10th minutes after the heel puncture
Change in oxygen saturation from 3rd minute before the heel puncture to 10th minute after the heel puncture | Measure the oxygen saturation at 10th minute after the heel puncture
  Measure the oxygen saturation at 3rd minute before the heel puncture, during, and at 1st, 5th and 10th minutes after the heel puncture

SECONDARY OUTCOMES:
Change in respond of pain from 3rd minute before the heel puncture to 10th minute after the heel puncture | Measure the NIPS at 3rd minute before the heel puncture
  Pain response assessed using the Neonatal Infants Pain Scale (NIPS), The evaluation indicators include 6 behavior indicators: facial expression, crying, breathing pattern, arms, legs and awakening status, except that the crying score is divided into three points (0, 1, 2 points), and the rest are two points (0 , 1 point), the total score is 0-7 points, the higher the score, the more serious the pain.
Change in respond of pain from 3rd minute before the heel puncture to 10th minute after the heel puncture | Measure the NIPS during the heel puncture
  Pain response assessed using the Neonatal Infants Pain Scale (NIPS), The evaluation indicators include 6 behavior indicators: facial expression, crying, breathing pattern, arms, legs and awakening status, except that the crying score is divided into three points (0, 1, 2 points), and the rest are two points (0 , 1 point), the total score is 0-7 points, the higher the score, the more serious the pain.
Change in respond of pain from 3rd minute before the heel puncture to 10th minute after the heel puncture | Measure the NIPS at 1st minute after the heel puncture
  Pain response assessed using the Neonatal Infants Pain Scale (NIPS), The evaluation indicators include 6 behavior indicators: facial expression, crying, breathing pattern, arms, legs and awakening status, except that the crying score is divided into three points (0, 1, 2 points), and the rest are two points (0 , 1 point), the total score is 0-7 points, the higher the score, the more serious the pain.
Change in respond of pain from 3rd minute before the heel puncture to 10th minute after the heel puncture | Measure the NIPS at 5th minute after the heel puncture
  Pain response assessed using the Neonatal Infants Pain Scale (NIPS), The evaluation indicators include 6 behavior indicators: facial expression, crying, breathing pattern, arms, legs and awakening status, except that the crying score is divided into three points (0, 1, 2 points), and the rest are two points (0 , 1 point), the total score is 0-7 points, the higher the score, the more serious the pain.
Change in respond of pain from 3rd minute before the heel puncture to 10th minute after the heel puncture | Measure the NIPS at 10th minute after the heel puncture
  Pain response assessed using the Neonatal Infants Pain Scale (NIPS), The evaluation indicators include 6 behavior indicators: facial expression, crying, breathing pattern, arms, legs and awakening status, except that the crying score is divided into three points (0, 1, 2 points), and the rest are two points (0 , 1 point), the total score is 0-7 points, the higher the score, the more serious the pain.

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang-Ming University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alemdar DK, Ozdemir FK. Effects of Covering the Eyes versus Playing Intrauterine Sounds on Premature Infants' Pain and Physiological Parameters during Venipuncture. J Pediatr Nurs. 2017 Nov-Dec;37:e30-e36. doi: 10.1016/j.pedn.2017.06.016. Epub 2017 Jul 24. PMID 28751136
- [Background] Alemdar DK. Effect of recorded maternal voice, breast milk odor, and incubator cover on pain and comfort during peripheral cannulation in preterm infants. Appl Nurs Res. 2018 Apr;40:1-6. doi: 10.1016/j.apnr.2017.12.001. Epub 2017 Dec 14. PMID 29579482
- [Background] Carvalho MES, Justo JMRM, Gratier M, Tome T, Pereira E, Rodrigues H. Vocal responsiveness of preterm infants to maternal infant-directed speaking and singing during skin-to-skin contact (Kangaroo Care) in the NICU. Infant Behav Dev. 2019 Nov;57:101332. doi: 10.1016/j.infbeh.2019.101332. Epub 2019 Aug 14. PMID 31421391
- [Background] Chirico G, Cabano R, Villa G, Bigogno A, Ardesi M, Dioni E. Randomised study showed that recorded maternal voices reduced pain in preterm infants undergoing heel lance procedures in a neonatal intensive care unit. Acta Paediatr. 2017 Oct;106(10):1564-1568. doi: 10.1111/apa.13944. Epub 2017 Jul 5. PMID 28580602
- [Background] Flacking R, Breili C, Eriksson M. Facilities for presence and provision of support to parents and significant others in neonatal units. Acta Paediatr. 2019 Dec;108(12):2186-2191. doi: 10.1111/apa.14948. Epub 2019 Sep 2. PMID 31350769